CLINICAL TRIAL: NCT00986960
Title: Effect of Pulsed ACTH add-on Therapy to Weekly Avonex on Remyelination and Neuroregeneration in Patients With Relapsing Remitting Multiple Sclerosis. A 1-year Placebo-controlled, Double-blinded, Randomized Follow-up Study
Brief Title: Effect of Adrenocorticotropin Injection With Weekly Interferon Beta in Patients With Relapsing Remitting Multiple Sclerosis (MS)
Acronym: ACTH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult to recruit due to protocol requirements - participant burden.
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NDA 08-372; NDA 08-372
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; relapsing remitting; RRMS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adrenocorticotropin hormone (Active Comparator): Patients receive the hormone
  Interventions: Drug: repository corticotropin injection
- Placebo (Placebo Comparator): Patients receive placebo only
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: repository corticotropin injection — IM ACTH: 80 units of Acthra gel I.M. once a day for 5 consecutive days at study time points 0, 3, 6, 9, and 12 months
  Other Names: H.P. Acthar gel
  Arms: Adrenocorticotropin hormone
Drug: Saline — I.M. placebo - 1ml of saline I.M. once per day for 5 consecutive days at 0, 3, 6, 9, and 12 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether the use of ACTH in addition to Avonex is effective in the treatment of relapsing remitting multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, immune-mediated disease of the central nervous system (CNS). It is a complex, multi-factorial disease that includes inflammatory and neurodegenerative processes manifesting both focally in the form of lesions and diffusely in otherwise normal-appearing brain tissue. Recent data shows that ACTH can have beneficial effects on specific neurodegenerative diseases and it may have superior neuroprotective effects. Adding a regimen of ACTH to standard Avonex treatment may provide neuroprotection and promote remyelination.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with MS according to McDonald criteria
* Age 18-65
* Have a RR disease course
* Have EDSS scores 0-5.5
* Have a disease duration <20 years
* Sub-optimal response to Interferon beta-1a I.M. (Avonex®) while being on therapy for at least 6 months defined as:
* presence of a documented relapse within the last 12 months
* or the presence of at least one enhancing T1 Gd lesion on an MRI performed within previous 3 months
* Signed informed consent
* Normal kidney functioning (creatinine clearance >59)
* None of the exclusion criteria

Exclusion Criteria:

* Presence of relapse or steroid treatment within 60 days prior to study enrollment
* Presence of neutralizing antibodies to IFNβ-1a I.M. prior to study enrollment
* Presence of optic neuritis within less than 6 months prior to study enrollment
* Diagnosis of osteoporosis (T score ≥2.5 SD)
* Women who are pregnant, lactating or of childbearing age who do not consent to approved contraceptive use during the study.
* Abnormal blood tests, performed during the screening visit including: hepatitis B or hepatitis C, ALT or AST greater than two times the upper limit of normal, abnormal glucose fasting levels or already known diabetes
* History of depression while on IFNβ-1a I.M.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To define the effect of add-on pulsed IM ACTH vs. placebo to IFNβ-1a I.M. on a voxel-wise MTR dynamic mapping of the lesions and NABT in patients with RRMS | 1 year
  Effect of ACTH in MRI

SECONDARY OUTCOMES:
To define the effect of add-on pulsed IM ACTH vs. placebo to IFNβ-1a I.M. in RRMS on anterior optic pathway pathology, as measured by OCT and LCLA in patients with RRMS. | 1 year
  Effect of ACTH on optic health

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — Buffalo Neuroimaging Analysis Center; Bianca Weinstock-Guttman, MD, Principal Investigator — Jacobs Neurological Institute
Locations (1):
- University at Buffalo, Buffalo General Hospital, Buffalo, New York, United States